CLINICAL TRIAL: NCT05607108
Title: Phase 2 Trial of ZEN003694 in Squamous Cell Lung Cancer Patients Harboring NSD3 Amplification
Brief Title: A Study of ZEN003694 in People With Squamous Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Zenith Epigenetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-286
Record Dates: First submitted 2022-11-01; First posted 2022-11-07 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Squamous Cell Lung Cancer
Keywords: Metastatic; Recurrent; ZEN003694; NSD3 Amplification; 22-286
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence

STUDY DESIGN:
Intervention Model Description: This is a single-arm phase 2 study of ZEN003694 in patients with advanced NSD3- amplified squamous cell lung cancer.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZEN003694 (Experimental): All patients enrolled on the study will undergo treatment with ZEN003694 60mg po qd on a 5 days on/2 days off schedule in an every 21-day cycle. All assessments, including drug dosing, have a window of +/- 7 days unless otherwise noted.
  Interventions: Drug: ZEN003694

INTERVENTIONS:
Drug: ZEN003694 — ZEN003694 60mg po qd on a 5 days on 2 days off schedule in an every 21-day cycle

SUMMARY:
The purpose of this study is to find out whether ZEN003694 is an effective treatment for people with advanced squamous cell lung cancer with a mutation in the NSD3 gene.

ZEN003694 is a type of drug called a BET inhibitor. Researchers think ZEN003694 may help here because the drug works by blocking a group of proteins called bromodomain and extra-terminal (BET) proteins, which may counteract the effect of NSD3 on tumor growth. Blocking these proteins may slow or stop the growth of the cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed squamous cell lung cancer
* Recurrent or metastatic disease
* Patients with previously treated asymptomatic brain metastases requiring no more than 10mg prednisone (or equivalent) are allowed. Patients with asymptomatic brain metastases ≤ 1cm not requiring more than 10mg prednisone (or equivalent) are allowed.
* Received prior first-line therapy: platinum-based chemotherapy and immunotherapy, given either concurrently or sequentially
* Eastern Cooperative Oncology Group (ECOG) PS 0-2
* Evidence of NSD3 gain or amplification by NGS, including but not limited to evidence of 8p11 gain or amplification as determined by MSK IMPACT or MSK ACCESS, or a commercially available molecular assay that is FDA authorized. Note: ctDNA testing, including but not limited to MSK ACCESS and Guardant and Foundation
* Adequate laboratory parameters at Screening including:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
  * Platelet count ≥ 100,000/mm^3
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.0 ULN (≤ 5 x ULN if liver metastases are present)
  * Total bilirubin ≤ 1.25 x ULN
  * Calculated or measured eGFR ≥ 40 ml/min or serum creatinine ≤ 1.5 x ULN
  * Prothrombin time (PT), international normalized ratio (INR) and partial thromboplastin time (PTT) < 1.5 x ULN
* Ability to swallow capsules
* Use of corticosteroids is allowed up to a daily dose of 10 mg prednisone or equivalent provided that the dose has been stable for at least 2 weeks prior to the start of ZEN003694 dosing and will remain stable during ZEN003694 treatment.
* Females or males age ≥ 18 years (at time of signing informed consent)
* Female subjects may be enrolled if they are not of childbearing potential, permanently sterile or who are post-menopausal defined as no menses for at least 1 year without an alternative medical cause and FSH levels in the post-menopausal range. Female subjects of childbearing potential may be enrolled if they consistently and correctly use a highly effective form of contraception. Highly effective forms of contraception include: combined (estrogen and progestogen hormonal contraceptives (oral, intravaginal, transdermal) associated with inhibition of ovulation; progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomized partner; sexual abstinence. Female subjects should not donate eggs from the time point of study drug administration until at least 7 months thereafter.
* Males with partners of childbearing potential may be enrolled if they use a condom when having sex with a pregnant woman or with a non-pregnant female of childbearing potential from 21 days before the first dose of study drug through 4 months after the last dose of study drug, and males should not donate sperm from the time point of study drug administration until at least 4 months thereafter.

Contraception should be considered for a non-pregnant female partner of childbearing potential

* Females of childbearing potential must have a negative serum or urine pregnancy test before the first dose of study drugs and must agree to pregnancy tests during the study.
* Females may not be breast-feeding at the first dose of study drugs, during study participation or through 7 months after the last dose of study drugs

Exclusion Criteria:

* Have previously received an investigational BET inhibitor
* Have received prior systemic anti-cancer therapy or investigational therapy within 2 weeks or five half-lives, whichever is shorter, prior to the first dose of study drug
* Radiation therapy within 2 weeks of first dose of study drug
* Currently receiving medications known to be strong inducers or inhibitors of CYP3A4 and substrates of CYP1A2 with a narrow therapeutic window. Strong inducers and inhibitors of CYP3A4 and CYP1A2 substrates with narrow therapeutic ranges must be discontinued at least 7 days prior to the first administration of study drug.
* Left ventricular ejection fraction less than the lower of 50% or the lower limit of institution's normal range
* QTcF interval > 470 msec
* Known impaired cardiac function or clinically significant cardiac disease such as uncontrolled supraventricular arrhythmia, ventricular arrhythmia requiring therapy, or uncontrolled congestive heart failure (New York Heart Association functional class III or IV)
* Myocardial infarction or unstable angina within 6 months prior to the first administration of study drug
* Other clinically significant co-morbidities, such as uncontrolled pulmonary disease, active CNS disease, active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy, or any other condition that could compromise safety or the patient's participation in the study
* Other known active cancer requiring therapy at time of study entry
* Historically positive (screening tests not required) for human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) or with active infections. HBV positivity defined by positive hepatitis B surface antigen (HBsAg). HCV positivity defined as positive HCV viral load.
* Major surgery other than diagnostic surgery, dental surgery or stenting within 4 weeks prior to the first administration of study drug
* History of congenital or other deficiency in platelet function, or any known inherent or acquired coagulopathy, including current anticoagulation therapy (except for low-dose warfarin for port patency)
* Current or anticipated use within 7 days prior to the first administration of study drug, or during the study, of strong P-gp inhibitors.
* Use of oral Factor Xa inhibitors (i.e., rivaroxaban, apixaban, betrixaban, edoxaban otamixaban, letaxaban, eribaxaban) and Factor IIa inhibitors (i.e., dabigatran). Low molecular weight heparin is allowed. Note: except for subjects on anticoagulant therapy who must have PT-INR within therapeutic range as deemed appropriate by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) | 2 years
  Response to ZEN003694 will be determined using the sum unidimensional measurements of the target lesions present on the scan. Unidimensional measurement rules will adhere to RECIST 1.1 guidelines.(6) Classification of response will be categorized by RECIST 1.1 (CR, PR, SD, PD).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Paik, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge Limited Protocol Activities, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (All Protocol Activities ), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm